CLINICAL TRIAL: NCT07291570
Title: Precision Detection and Prediction of Atrial Arrhythmias Using Artificial Intelligence and Consumer Wearable Devices (REMOTE-AF2)
Brief Title: Precision Detection and Prediction of Atrial Arrhythmias Using Artificial Intelligence and Consumer Wearable Devices
Acronym: REMOTE-AF2
Status: Not yet recruiting | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 354811; C0118: RFSG-26/2 (Other Grant/Funding Number: Royal Brompton and Harefield Hospitals Charity)
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-10

CONDITIONS: Atrial Fibrillation (AF)
Keywords: atrial fibrillation; remote monitoring; artificial intelligence; wearables; photophlethysmography (PPG)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Wearable

SUMMARY:
Atrial fibrillation (AF) is the most prevalent cardiac arrhythmia affecting over one million people in the UK. It is associated with increased cardiovascular morbidity and mortality and costs the NHS between £1.4 billion and 2.5 billion annually. Current methods to detect AF include opportunistic pulse palpation, single time point 12-lead electrocardiograms (ECGs), ambulatory Holter monitoring, and implantable loop recorders (ILRs). The more widely used intermittent monitoring methods, such as ECGs and Holter monitoring, are limited in terms of duration and have lower detection yields of atrial arrhythmias. At the other end of the spectrum, the ILR can give continuous and accurate arrhythmia detection but is invasive and requires specialist expertise to implant, monitor, and analyse.

In recent years, the use of wearable mobile health (mHealth) devices has emerged as a direct-to-consumer option for monitoring parameters such as heart rate and activity levels. From a clinical perspective they potentially offer a less invasive and cost-effective investigative approach, with remote monitoring solutions to possibly predict and detect AF. This technology has significant potential in terms of passive, non-invasive and continuous monitoring to aid the early diagnosis and management of AF.

The original REMOTE-AF study (NCT05037136) developed novel methodology to detect AF using PPG-dervived data from a wearable. This study will further enhance this foundational work by recruiting patients to develop a AI-enabled, multi-parametric algorithm using PPG-derived data to detect AF.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 and above with a confirmed diagnosis of paroxysmal AF or those who have undergone treatment for paroxysmal, or persistent AF and had sinus rhythm restored.
2. Capability to provide informed consent, coupled with self-reported sufficiency of digital literacy.
3. Regular access to a Wi-Fi connection (at least weekly).
4. Own a smartphone (released after 2017).

Exclusion Criteria:

1. Individuals with permanent or persistent AF that remains uncontrolled despite receiving treatment.
2. Conditions or disabilities that preclude adherence to study instructions or proper use of the devices.
3. A known severe allergy to any of the materials in the wearable or ECG device poses a risk to participant safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed diagnosis of paroxysmal AF or persistent AF who have undergone treatment to restore sinus rhythm
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
To evaluate the accuracy of an AI algorithm based on PPG-derived metrics in predicting and detecting AF against intermittent rhythm monitoring. | 6 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Brompton and Harefield Hospitals, Guy's and St Thomas' NHS Foundation Trust, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adasuriya G, Barsky A, Kralj-Hans I, Mohan S, Gill S, Chen Z, Jarman J, Jones D, Valli H, Gkoutos GV, Markides V, Hussain W, Wong T, Kotecha D, Haldar S. Remote monitoring of atrial fibrillation recurrence using mHealth technology (REMOTE-AF). Eur Heart J Digit Health. 2024 Feb 12;5(3):344-355. doi: 10.1093/ehjdh/ztae011. eCollection 2024 May. PMID 38774381